CLINICAL TRIAL: NCT01274065
Title: Developing an Interdisciplinary Pharmacogenomic Treatment Approach to Reduce Medication Burden and Improve Subject Outcomes
Brief Title: Developing an Interdisciplinary Pharmacogenomic Treatment Approach to Reduce Medication Burden and Improve Outcomes
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: ARI-1290-Pharm
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Developmental Disabilities
Keywords: psychiatry; psychiatric illness; developmental disability; mental health; medication burden
MeSH Terms: conditions — Developmental Disabilities; Mental Disorders; Psychological Well-Being | interventions — Genetic Testing; Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psychiatric illnesses: Participants will reside at the South Dakota Developmental Center (SDDC), which serves a unique population of people with developmental disabilities and co-occuring psychiatric disorders.
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — The research team will review data following DNA sample analysis and identify variants in genes that result in impaired drug metabolism
  Other Names: pharmacogenomics

SUMMARY:
There is no common rule as to how a drug will affect patients. This is due to the effect specific DNA sequences of genes have on drug response, by the effect they have on how medications are metabolized. The primary objective of this research is to optimize medication therapy and to reduce the number of medications used, specifically medications for people with developmental disabilities and co-occuring psychiatric illnesses.

DETAILED DESCRIPTION:
The primary goal of this study is to develop a process for utilizing pharmacogenomic analysis as a strategy to improve the quality of life, safety, decrease medication burden, and enhance the effectiveness of medications in people with psychiatric illnesses and developmental disabilities. Ultimately, this inter-disciplinary service could be developed into a standard screening and consultation tool for healthcare providers to utilize when determining the most appropriate medication for their patients.

ELIGIBILITY:
Inclusion Criteria:

* Current resident of the South Dakota Developmental Center (SDDC)
* Currently taking a high number of medications per month
* Eligibility of the subjects will be determined by the treatment team which consists of 3-4 of the following individuals: treating psychologist, behavior therapist, case manager, supervisors, counselors, dietitians, physician assistants, occupational therapists, and physical therapists

Exclusion Criteria:

* To be determined by the research staff

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study participants will all reside at the South Dakota Developmental Center (SDDC), which serves a unique population of people with developmental diabilities and co-occuring psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Soundy, MD, Principal Investigator — Avera McKennan Hospital & University Health Center

REFERENCES:
- [Background] Zhou SF, Di YM, Chan E, Du YM, Chow VD, Xue CC, Lai X, Wang JC, Li CG, Tian M, Duan W. Clinical pharmacogenetics and potential application in personalized medicine. Curr Drug Metab. 2008 Oct;9(8):738-84. doi: 10.2174/138920008786049302. PMID 18855611
- [Background] Oscarson M. Pharmacogenetics of drug metabolising enzymes: importance for personalised medicine. Clin Chem Lab Med. 2003 Apr;41(4):573-80. doi: 10.1515/CCLM.2003.087. PMID 12747605
- [Background] Deeken J. The Affymetrix DMET platform and pharmacogenetics in drug development. Curr Opin Mol Ther. 2009 Jun;11(3):260-8. PMID 19479659
- [Background] de Leon J, Armstrong SC, Cozza KL. Clinical guidelines for psychiatrists for the use of pharmacogenetic testing for CYP450 2D6 and CYP450 2C19. Psychosomatics. 2006 Jan-Feb;47(1):75-85. doi: 10.1176/appi.psy.47.1.75. PMID 16384813